CLINICAL TRIAL: NCT01511510
Title: A Phase I, Randomized, Subject And Investigator Blind, Sponsor Open, Multiple Escalating Dose Study To Evaluate The Safety, Tolerability And Pharmacokinetics Of PF-04958242 In Healthy Adult Volunteers
Brief Title: Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Repeated Doses of PF-04958242 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B1701007
Record Dates: First submitted 2011-07-19; First posted 2012-01-18 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Schizophrenia
Keywords: PF-04958242; multiple dose; safety; schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — PF-04958242

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04958242 (Experimental)
  Interventions: Drug: PF-04958242
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04958242 — PF-04958242 0.05 mg oral solution Q24 hours for 14 days
  Arms: PF-04958242
Drug: PF-04958242 — PF-04958242 0.10 mg oral solution Q24 hours for 14 days
  Arms: PF-04958242
Drug: PF-04958242 — PF-04958242 0.15 mg oral solution Q24 hours for 14 days
  Arms: PF-04958242
Drug: PF-04958242 — PF-04958242 0.25 mg oral solution Q24 hours for 14 days
  Arms: PF-04958242
Drug: Placebo — Placebo oral solution Q24 hours for 14 days
  Arms: Placebo

SUMMARY:
This study aims to assess the safety, tolerability, and pharmacokinetics of PF-04958242 at a number of ascending doses administered once daily for 14 days in healthy volunteers.

DETAILED DESCRIPTION:
This study was previously posted by Pfizer, Inc. Sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-child bearing potential Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs)

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease
* History of seizures or of a condition with risk of seizures
* Pregnant or nursing females, and females of child bearing potential

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Composite of Pharmacokinetics measured at 0.25, 0.5, 0.75, 1, 2, 3, 4, 8, 12, 24 hours after dosing on Day 1 | Day 1-Day 2
Composite of Pharmacokinetics measured pre-dose and 1 hour post-dose on Day 4 | Day 4
Composite of Pharmacokinetics measured pre-dose and 1 hour post-dose on Day 7 | Day 7
Composite of Pharmacokinetics measured at 0.25, 0.5, 0.75, 1, 2, 3, 4, 8, 12, 24, 48, 72, 120 hours after dosing on Day 14 | Day 14-Day 18
Composite of urine Pharmacokinetics measured for 24 hours post-dose on Day 14 | Day 14-Day 15

SECONDARY OUTCOMES:
Drug Effect Questionaire Liking scale | Day 14
Digit Symbol Substitution Test | Day 14
Columbia Suicide Severity Rating Scale | Day 0-Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1701007&StudyName=Study%20to%20Evaluate%20the%20Safety%2C%20Tolerability%20and%20Pharmacokinetics%20of%20Repeated%20Doses%20of%20PF-04958242%20in%20Healthy%20Volunteers%20